CLINICAL TRIAL: NCT01928719
Title: Reduced Nicotine Content Cigarettes in Smokers of Lower Socioeconomic Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: George Washington University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 43804UG-P1; P50DA036107-01 (NIH)
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Tobacco Dependence
Keywords: Smoking; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Nicotine Content Cigarettes (Experimental): the experimental group will smoke cigarettes with Gradually Reduced Nicotine Content (RNC) (11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg per cigarette) cigarettes, each smoked for 3 weeks, except for the last period which will last 6 weeks to evaluate a longer-term adherence to the lowest nicotine content cigarette.
  Interventions: Drug: Reduced Nicotine Content Cigarettes
- Same Nicotine Content Cigarettes (Placebo Comparator): The Same Nicotine Control Group (SNC) will continue to smoke research cigarettes with a usual nicotine content (about 11.6 mg per cigarette)
  Interventions: Drug: Same Nicotine Content Cigarettes

INTERVENTIONS:
Drug: Reduced Nicotine Content Cigarettes — Cigarettes contain 11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg nicotine per cigarette
  Other Names: Nicotine
  Arms: Reduced Nicotine Content Cigarettes
Drug: Same Nicotine Content Cigarettes — about 11.6 mg nicotine per cigarette
  Other Names: Nicotine
  Arms: Same Nicotine Content Cigarettes

SUMMARY:
The overall goal of this study is to address the question of whether progressively lowering nicotine content in cigarettes can reduce or eliminate nicotine dependence in smokers of low socioeconomic status

DETAILED DESCRIPTION:
To address the question of whether progressively lowering nicotine content in cigarettes can reduce or eliminate nicotine dependence in low socioeconomic smokers, we will randomize smokers to either an Reduced Nicotine Content group with a gradual step-wise reduction in nicotine from 11 mg to 0.2 mg per cigarette in five 3-wk stages, or a control group with nicotine content similar to their preferred usual brand of cigarettes.

Overall, we hypothesize that low socioeconomic smokers who switch to progressively lower nicotine cigarettes will initially alter their smoking behavior to compensate for lower nicotine until cigarette nicotine yields become so low that complete compensation becomes too difficult. At that point, smokers will either drop-out or continue to smoke the reduced nicotine content cigarettes but with incomplete compensatory behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Less than 16 years of education
* Able to understand, and sign consent
* Smoke >4 cigarettes/day for at least a year
* No quit attempt in prior 1 month and not planning to quit smoking within next 6 months
* Plan to live in local area for next 8 months
* Able to read and write in English
* Women not pregnant and taking steps to avoid pregnancy

Exclusion Criteria:

* College graduate
* Use of psychotropic drugs
* Significant medical condition, or immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data
* Use of any non-cigarette nicotine delivery product in the past week or smoking cessation medicine in prior 3 months
* Currently pregnant or nursing
* Uncontrolled serious psychotic illness or substance abuse
* History of difficulties providing blood samples-fainting, poor veins, anxiety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Muscat, PhD, Principal Investigator — Penn State College of Medicine; Kimberly Horn, PhD, Study Director — George Washington University School of Public Health
Locations (2):
- United States (2):
  - George Washington University School of Public Health, Washington D.C., District of Columbia
  - Penn State College of Medicine, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krebs NM, Allen SI, Veldheer S, Martinez DJ, Horn K, Livelsberger C, Modesto J, Kuprewicz R, Wilhelm A, Hrabovsky S, Kazi A, Fazzi A, Liao J, Zhu J, Wasserman E, Reilly SM, Reinhart L, Trushin N, Moyer RE, Bascom R, Foulds J, Richie JP Jr, Muscat JE. Reduced nicotine content cigarettes in smokers of low socioeconomic status: study protocol for a randomized control trial. Trials. 2017 Jul 3;18(1):300. doi: 10.1186/s13063-017-2038-9. PMID 28673312

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a baseline phase of one week on usual brand cigarettes and another baseline phase on same nicotine content cigarettes (2 weeks). Of these, 35 participants either were lost to follow up or withdrawn from the study during the baseline phase and before they started the intervention.
Groups:
- Reduced Nicotine Content Cigarettes: The experimental group will smoke cigarettes with Gradually Reduced Nicotine Content (RNC) (11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg per cigarette) cigarettes, each smoked for 3 weeks, except for the last period which will last 6 weeks to evaluate a longer-term adherence to the lowest nicotine content cigarette. Cigarettes contain 11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg nicotine per cigarette
Period: Overall Study
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Started | 122 | 123
Completed | 70 | 104
Not Completed | 52 | 19
Not completed — Lost to Follow-up | 26 | 11
Not completed — Withdrawal by Subject | 22 | 7
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline values for outcomes reflect levels after participants were on the usual nicotine content cigarettes for 2 weeks and before they received the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (12.1) | 45.1 (10.8) | 44.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 72 | 128
  Male | 66 | 51 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 117 | 120 | 237
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/white | 71 | 82 | 153
  African American/black | 43 | 35 | 78
  Asian | 1 | 0 | 1
  Native Hawaiian or Pacific Island | 1 | 1 | 2
  American Indian/Alaskan native | 0 | 3 | 3
  Other | 5 | 1 | 6
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 122 | 123 | 245
Education [Count of Participants; unit: Participants]
  < High School Degree | 15 | 25 | 40
  High School Degree | 55 | 57 | 112
  > High School Degree and < Bachelor's degree | 52 | 41 | 93
Cigarettes per Day [Mean (Standard Deviation); unit: cigarettes] | 24.2 (11) | 24 (13.9) | 24.1 (12.5)
Plasma Cotinine [Mean (Standard Deviation); unit: ng/ml] — Samples below the level of detection were set to 3 ng/mL.
  ng/ml | 261.6 (148.6) | 260.3 (148.5) | 260.9 (148.3)
Exhaled Carbon Monoxide [Mean (Standard Deviation); unit: parts per million] | 31.5 (17.2) | 31.3 (15.8) | 31.4 (16.5)
Perceived Stress Scale Score [Mean (Standard Deviation); unit: units on a scale] — 10-item version was used. Scale range is 0-40. Higher scores indicate more stress.
  units on a scale | 12.6 (6.7) | 12.1 (7.2) | 12.3 (6.9)
Menthol smoker [Count of Participants; unit: Participants] | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Dropped Out of Study as a Measure of Adherence
Description: Adherence to the regimen was assessed via dropout (due to withdrawal or lost-to-follow up) during the randomized intervention trial phase of the study. Dropout was analyzed as a time-to-event outcome during the 18 weeks after randomization.
Time Frame: 18 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 122 | 123
Participants | 52 | 19
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 3.3, 95% CI 2-sided [1.95 to 5.58] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

2. Secondary Outcome: Predictors of Participant Dropout
Description: Baseline participant characteristics were evaluated for their association with the primary outcome, randomized trial phase dropout. The table below reports the number of participants who dropped out by each characteristic that was found to be univariately associated with the primary outcome.
Time Frame: 18 weeks
Population: Participants (who were randomized) are stratified according to the listed characteristics.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The experimental group will smoke cigarettes with Gradually Reduced Nicotine Content (RNC) (11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg per cigarette) cigarettes, each smoked for 3 weeks, except for the last period which will last 6 weeks to evaluate a longer-term adherence to the lowest nicotine content cigarette. Cigarettes contain 11.6, 7.4, 3.3, 1.4, 0.7, and 0.2 mg nicotine per cigarette.
  The Same Nicotine Control Group (SNC) will continue to smoke research cigarettes with a usual nicotine content (about 11.6 mg per cigarette).
Arm/Group | All Participants
Number analyzed (Participants) | 245
Participants
  Reduced Nicotine Content Group: number analyzed (Participants) | 122
  Reduced Nicotine Content Group | 52
  Same Nicotine Content Group: number analyzed (Participants) | 123
  Same Nicotine Content Group | 19
  Age group 18-29: number analyzed (Participants) | 33
  Age group 18-29 | 20
  Age group 30-39: number analyzed (Participants) | 38
  Age group 30-39 | 14
  Age group 40-49: number analyzed (Participants) | 77
  Age group 40-49 | 15
  Age group 50-59: number analyzed (Participants) | 81
  Age group 50-59 | 18
  Age group 60-65: number analyzed (Participants) | 16
  Age group 60-65 | 4
  Not currently working: number analyzed (Participants) | 135
  Not currently working | 31
  Currently working: number analyzed (Participants) | 108
  Currently working | 40
  BMI Underweight (<18.5): number analyzed (Participants) | 9
  BMI Underweight (<18.5) | 6
  BMI Normal weight (>=18.5 and <25): number analyzed (Participants) | 63
  BMI Normal weight (>=18.5 and <25) | 17
  BMI Overweight (>=25 and <30): number analyzed (Participants) | 59
  BMI Overweight (>=25 and <30) | 15
  BMI Obese (>=30): number analyzed (Participants) | 114
  BMI Obese (>=30) | 33
Statistical Analysis 1: Comparison: All Participants; The reference group is Same Nicotine Content Group; Test type: Other; p < 0.0001, Regression, Cox — Testing the effect of treatment group in a Multivariable Cox Regression Model; Adjusting for Age Group, Working Status, and BMI; Hazard Ratio (HR) = 3.4, 95% CI 2-sided [1.99 to 5.81] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes
Statistical Analysis 2: Comparison: All Participants; The reference group is Age equals 18-29; Test type: Other; p = 0.06, Regression, Cox — Testing the effect of age group (ages 30-39) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and BMI; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.26 to 1.03] — The direction of comparison is Age group 30-39 to the Age group 18-29
Statistical Analysis 3: Comparison: All Participants; The reference group is Age equals 18-29; Test type: Other; p < 0.002, Regression, Cox — Testing the effect of age group (ages 40-49) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and BMI; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.17 to 0.66] — The direction of comparison is Age group 40-49 to the Age group 18-29
Statistical Analysis 4: Comparison: All Participants; The reference group is Age equals 18-29; Test type: Other; p < 0.002, Regression, Cox — Testing the effect of age group (Ages 50-59) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and BMI; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.16 to 0.65] — The direction of comparison is Age group 50-59 to Age group 18-29
Statistical Analysis 5: Comparison: All Participants; The reference group is Age equals 18-29; Test type: Other; p = 0.1, Regression, Cox — Testing the effect of age group (Ages 60-65) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and BMI; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.13 to 1.18] — The direction of comparison is Age group 60-65 to the Age group 18-29
Statistical Analysis 6: Comparison: All Participants; The reference group is not currently working; Test type: Other; p = 0.1, Regression, Cox — Testing the effect of working status in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Age, and BMI; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.92 to 2.66]; The direction of comparison is currently working to not currently working
Statistical Analysis 7: Comparison: All Participants; The reference group is BMI Underweight (<18.5); Test type: Other; p = 0.006, Regression, Cox — Testing the effect of BMI Normal Weight group (>=18.5 & <25) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and Age; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.1 to 0.67] — The direction of comparison is Normal Weight (>=18.5 & <25) to Underweight (<18.5) group
Statistical Analysis 8: Comparison: All Participants; The reference group is BMI Underweight group (<18.5); Test type: Other; p = 0.034, Regression, Cox — Testing the effect of BMI Overweight group (>=25 & < 30) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and Age; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.13 to 0.92] — The direction of comparison is Overweight (>=25 & < 30) to Underweight (<18.5) group
Statistical Analysis 9: Comparison: All Participants; The reference group is BMI Underweight group (<18.5); Test type: Other; p = 0.011, Regression, Cox — Testing the effect of BMI Obese group (>=30) in a Multivariable Cox Regression Model; Adjusting for Treatment Group, Working Status, and Age; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.13 to 0.77] — The direction of comparison is Obese (>=30) to Underweight (<18.5) group

3. Secondary Outcome: Cigarettes Per Day
Description: Measured by self-reported cigarettes per day at in-person clinic visits using 6-day follow back
Time Frame: 18 weeks
Population: All randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: cigarettes per day
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 122 | 123
cigarettes per day | 21.0 [19.2 to 22.8] | 25.1 [23.6 to 26.6]
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p = 0.0006, Mixed Models Analysis; The model included time, group, and time-by-group interaction; treating baseline scores for outcomes as covariates; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-6.44 to -1.75] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

4. Secondary Outcome: Nicotine Exposure
Description: Measured by cotinine (ng/ml) measured in plasma
Time Frame: 18 weeks
Population: All randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 122 | 123
ng/ml | 128.6 [101.9 to 155.2] | 265.3 [242.6 to 287.9]
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p < .0001, Mixed Models Analysis; The model included time, group, and time-by-group interaction; treating baseline scores for outcomes as covariates; Least Squares Mean Difference = -136.7, 95% CI 2-sided [-171.7 to -101.7] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

5. Secondary Outcome: Smoke Exposure
Description: Measured in carbon monoxide levels by expired CO
Time Frame: 18 weeks
Population: All randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: parts per million (ppm)
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 122 | 123
parts per million (ppm) | 27.2 [24.4 to 30.0] | 31.2 [28.9 to 33.6]
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p = 0.0305, Mixed Models Analysis; The model included time, group, and time-by-group interaction; treating baseline scores for outcomes as covariates; Least Squares Mean Difference = -4.03, 95% CI 2-sided [-7.68 to -0.38] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

6. Secondary Outcome: Perceived Stress
Description: Perceived Stress is measured via the Perceived Stress Scale Score. The 10-item version was used. Scale range is 0-40. Higher scores indicate more stress.
Time Frame: 18 weeks
Population: All randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 122 | 123
score on a scale | 12.9 [11.8 to 14.1] | 11.1 [10.2 to 12.11]
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p = 0.0207, Mixed Models Analysis; The model included time, group, and time-by-group interaction; treating baseline scores for outcomes as covariates; Least Squares Mean Difference = 1.81, 95% CI 2-sided [0.28 to 3.33] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

7. Secondary Outcome: Cortisol
Description: Salivary Cortisol Cortisol is produced by the hypothalamic-pituitary-adrenal axis (HPA) axis in response to stress. Peak cortisol measures during the cortisol awakening response were used.
Time Frame: 15 weeks
Population: A subset of participants was randomly selected to complete the cortisol collection procedure and those who provided usable samples 1-3 were used in this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dl
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
Number analyzed (Participants) | 15 | 27
ng/dl | 0.32 [-0.02 to 0.67] | 0.48 [0.29 to 0.68]
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Same Nicotine Content Cigarettes; Test type: Other; p = 0.4191, Mixed Models Analysis; The model included time, group, and time-by-group interaction; treating baseline scores for outcomes as covariates; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-0.56 to 0.23] — The direction of comparison is reduced nicotine content vs. same nicotine content cigarettes

ADVERSE EVENTS:
Time Frame: 33 weeks
Description: Adverse events (AEs) were systematically collected at each study visit by asking participants about any changes in their physical or mental health or if they needed to seek immediate medical care at an emergency room or hospital.
Arm/Group | Reduced Nicotine Content Cigarettes | Same Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 1/122 | 1/123
Serious Adverse Events (participants affected / at risk) | 11/122 | 11/123
Other Adverse Events (participants affected / at risk) | 54/122 | 63/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Nicotine Content Cigarettes (N=122) | Same Nicotine Content Cigarettes (N=123)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hernia
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Diabetes
Pain (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0) — Psychiatric hospitalization
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Breast cancer diagnosis
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (3)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Nicotine Content Cigarettes (N=122) | Same Nicotine Content Cigarettes (N=123)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Depression (Psychiatric disorders) | 7 (7) | 10 (10)
Flu like symptoms (General disorders) | 8 (9) | 4 (4)
Hypertension (Vascular disorders) | 12 (12) | 10 (11)
Respiratory, thoracic, and mediastinal disorders- Other (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 13 (13)
Surgical and medical procedures - Other (Surgical and medical procedures) | 9 (9) | 13 (14)
Upper respiratory infection (Infections and infestations) | 20 (26) | 21 (23)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)

LIMITATIONS AND CAVEATS:
The sample size was not reached due to a shortage of study cigarette inventory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT01928719/Prot_SAP_001.pdf